CLINICAL TRIAL: NCT04797013
Title: A Phase 3, Multicentre,Open-label, Randomised Controlled, Non-inferiority Trial
Brief Title: Tenecteplase Reperfusion Therapy in Acute Ischemic Cerebrovascular Events-Ⅱ
Acronym: TRACEⅡ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: CSPC Mingfule Pharmaceutical (Guangzhou) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yongjun Wang, President of Beijing Tiantan Hospital, Capital Medical University, Director of Neurology Center, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MK02-2020-01
Record Dates: First submitted 2021-02-25; First posted 2021-03-15 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Acute Ischemic Stroke
Keywords: rhTNK-tPA; acute; stroke; phaseⅢ; Acute Ischemic Stroke; rt-PA
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Tissue Plasminogen Activator; Injections

STUDY DESIGN:
Intervention Model Description: multicenter, prospective, randomized, open label, blinded-endpoint (PROBE)，Parallel controls，Non-inferiority
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhTNK-tPA (0.25mg/kg) (Active Comparator): rhTNK-tPA (0.25mg/kg) is given as a single, intravenous bolus (within 5-10 seconds) immediately upon randomization. Maximum dose 25mg.
  Interventions: Drug: rhTNK-tPA
- rt-PA (0.9mg/kg) (Active Comparator): 10% dose of rt-PA (0.9 mg/kg) is given as bolus and the remainder in 1 hour. Maximum dose 90mg.
  Interventions: Drug: rt-PA

INTERVENTIONS:
Drug: rt-PA — Subjects will be randomized to rhTNK-tPA or rt-PA in a 1:1 ratio.
  Other Names: Alteplase injection (rt-PA)
  Arms: rt-PA (0.9mg/kg)
Drug: rhTNK-tPA — Subjects will be randomized to rhTNK-tPA or rt-PA in a 1:1 ratio.
  Other Names: Recombinant Human TNK Tissue-type Plasminogen Activator for Injection
  Arms: rhTNK-tPA (0.25mg/kg)

SUMMARY:
A Phase Ⅲ, Multicenter, Prospective, Randomized, Open Label, Blinded-endpoint (PROBE) Controlled Trial of Recombinant Human TNK Tissue-type Plasminogen Activator (rhTNK-tPA) for Injection Versus Alteplase for Acute Ischemic Stroke Within 4.5 Hours

DETAILED DESCRIPTION:
To test the hypothesis that rhTNK-tPA is non-inferior to alteplase in thrombolysis treatment when administered within 4.5 hours of ischemic stroke onset.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, no gender limitation;
* The time from onset to treatment was < 4.5h;The time at which symptoms begin is defined as "the time at which they finally appear normal";
* The clinical diagnosis was ischemic stroke (the diagnosis followed the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018);
* MRS before onset was 0-1 points
* Baseline NIHSS 5-25(both included);
* Informed consent from the patient or surrogate.

Exclusion Criteria:

* Intended to proceed endovascular treatment;
* NIHSS consciousness score >2;
* Allergy to tenecteplase or alteplase;
* Past history of intracranial hemorrhage ;
* A history of severe head trauma or stroke within 3 months;
* A history of intracranial or spinal surgery within 3 months;
* A history of gastrointestinal or urinary bleeding within 3 weeks;
* 2 weeks of major surgery;
* Arterial puncture was performed at the hemostasis site that was not easily compressed within 1 week;
* Intracranial tumors (except neuroectodermal tumors, such as meningiomas), large intracranial aneurysms;
* Intracranial hemorrhage (including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, subdural/extradural hematoma, etc.);
* Active visceral bleeding;
* Aortic arch dissection was found;
* After active antihypertensive treatment, hypertension is still not under control: systolic blood pressure ≥180 mm Hg, or diastolic blood pressure ≥100 mm Hg;
* Propensity for acute bleeding, including platelet counts of less than 100×109/ L or otherwise;
* Blood glucose <2.8 mmol/L or >22.22 mmol/L;
* Oral warfarin anticoagulant with INR>1.7 or PT>15 s;
* Heparin treatment was received within 24 h;
* Thrombin inhibitors or factor Xa inhibitors were used within 48 h;
* Head CT or MRI showed a large infarction (infarcted area > 1/3 of the middle cerebral artery);
* Subjects who are unable or unwilling to cooperate due to hemiplegia (Todd's palsy) after epileptic seizure or other neurological/psychiatric disorders;
* Pregnant women, lactating women, or subjects who do not agree to use effective contraception during the trial;
* Participation in other clinical trials within 3 months prior to screening;
* Unsuitability or participation in this study as judged by the Investigator may result in subjects being exposed to greater risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1430 (Actual)
Dates: Start 2021-06-12 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Excellent functional outcome | 90 days
  Proportion of subjects with mRS(0-1) at 90 days.

SECONDARY OUTCOMES:
Good functional outcome | 90 days
  Proportion of subjects with mRS(0-2) at 90 days.
National Institutes of Health Stroke Scale (NIHSS) | 24 hours，day7
  Proportion of subjects with NIHSS score ≥ 4 improved compared with baseline at 24 or with NIHSS 0-1 at 24 hours and 7 days.
EQ-5D | 90 days
  Quality of life measured by EQ-5D scale.
Barthel (BI) | 90 days
  Global function of daily living defined as BI ≥ 95 at 90 days.
Modified Rankin Scale(mRS) | 90 days
  Ordinal distribution of mRS at 90 days.

OTHER OUTCOMES:
Symptomatic intracranial hemorrhage(sICH) | 36 hours
  Proportion of subjects with symptomatic intracranial hemorrhage (sICH) at 36 hours.( defined by ECASSIII)
Asymptomatic intracranial hemorrhage | 90 days
  The incidence of asymptomatic intracranial hemorrhage at 90 days.
PH2 intracranial hemorrhage | 90 days
  The incidence of PH2 intracranial hemorrhage within 90 days (according to SITS standards).
Any intracranial hemorrhage | 90 days
  The incidence of any intracranial hemorrhage within 90 days.
Systematic bleeding | 90 days
  The incidence of Systematic bleeding at 90 days.( defined by GUSTO）
Deaths | 90 days
  Rate of Overall mortality at 90 days.
AEs/SAEs | 90 days
  The incidence of adverse events(AEs) / severe adverse events(SAEs) at 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Sun, Study Director — IRB of Beijing Tiantan Hospital,Capital Medical University
Locations (61):
- China (61):
  - The first affiliated hospital of ustc, Hefei, Anhui
  - The people's hospltal of xuancheng city, Xuancheng, Anhui
  - Beijing luhe hospital capital medical university, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - The first hospital of lanzhou university, Lanzhou, Gansu
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangdong, Guangdong
  - Yue bei people's hospital, Shaoguan, Guangdong
  - Guizhou provincial people's hospital, Guiyang, Guizhou
  - Affiliated hospital of chengde medical university, Chengde, Hebei
  - The first hospital of hebei medical university, Shijiazhuang, Hebei
  - the Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan Workers ' Hospital, Tangshan, Hebei
  - The first affiliated hospital of hebei north university, Zhangjiakou, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The 2ad affiliated hospital of harbin medical university, Haerbin, Heilongjiang
  - Second People's Hospital of Jiaozuo City, Jiaozuo, Henan
  - Nanyang central hospital, Nanyang, Henan
  - Nanyang Nanshi Hospital, Nanyang, Henan
  - Nayang second general hospital, Nanyang, Henan
  - Pingmei Shenma Medical Group General Hospital, Pingdingshan, Henan
  - Xinxiang first people's hospital, Xinxiang, Henan
  - Xinyang central hospital, Xinyang, Henan
  - The first affiliated hospital of zhengzhou university, Zhengzhou, Henan
  - The central hospital of wuhan, Wuhan, Hunan
  - Inner Mongolia Baotou Hospita, Baotou, Inner Mongolia
  - Affiliated Hospital of Chifeng University, Chifeng, Inner Mongolia
  - Kashkten Mongolian Medicine Hospital, Chifeng, Inner Mongolia
  - Inner Mongolia People'S Hospital, Hohhot, Inner Mongolia
  - Huai an second people's hospital, Huaian, Jiangsu
  - Jiangsu taizhou people's hopital, Taizhou, Jiangsu
  - General Hospital of Xuzhou Mining Group, Xuzhou, Jiangsu
  - Xuzhou central hospital, Xuzhou, Jiangsu
  - Third Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - Jilin neuropsychiaric hospital, Siping, Jilin
  - Tonghua Central Hospital, Tonghua, Jilin
  - Meihekou Central Hospital, Tonghua, Jilin
  - The Firet Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Central hospital affiliated to shenyang medical college, Shenyang, Liaoning
  - General Hospital of Northern War Zone, PLA, Shenyang, Liaoning
  - The first hospital of china medical university, Shenyang, Liaoning
  - The First People'S Hospital of Shenyang, Shenyang, Liaoning
  - Linyi City People Hospital, Linyi, Shandong
  - Tengzhou Central People's Hospital, Tengzhou, Shandong
  - Yantai Yuhuangding Hosopital, Yantai, Shandong
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Heping hospital affiliated to changzhi medical college, Changzhi, Shanxi
  - General Hospital of Chinese Medicine and Coal, Datong, Shanxi
  - The fifth people's s hospital of datong, Datong, Shanxi
  - Linfen central hospital, Linfen, Shanxi
  - Linfen people's hospital, Linfen, Shanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - Xianyang Hospital of Yan ' an University, Xianyang, Shanxi
  - Mianyang central hospital, Mianyang, Sichuan
  - Shanxi provincial prople's hospital, Taiyuan, Taiyuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang
  - Taizhou Enze Medical Center ( Group ), Taizhou, Zhejiang
  - Wenzhou Central Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell BCV, Mitchell PJ, Churilov L, Yassi N, Kleinig TJ, Dowling RJ, Yan B, Bush SJ, Thijs V, Scroop R, Simpson M, Brooks M, Asadi H, Wu TY, Shah DG, Wijeratne T, Zhao H, Alemseged F, Ng F, Bailey P, Rice H, de Villiers L, Dewey HM, Choi PMC, Brown H, Redmond K, Leggett D, Fink JN, Collecutt W, Kraemer T, Krause M, Cordato D, Field D, Ma H, O'Brien B, Clissold B, Miteff F, Clissold A, Cloud GC, Bolitho LE, Bonavia L, Bhattacharya A, Wright A, Mamun A, O'Rourke F, Worthington J, Wong AA, Levi CR, Bladin CF, Sharma G, Desmond PM, Parsons MW, Donnan GA, Davis SM; EXTEND-IA TNK Part 2 investigators. Effect of Intravenous Tenecteplase Dose on Cerebral Reperfusion Before Thrombectomy in Patients With Large Vessel Occlusion Ischemic Stroke: The EXTEND-IA TNK Part 2 Randomized Clinical Trial. JAMA. 2020 Apr 7;323(13):1257-1265. doi: 10.1001/jama.2020.1511. PMID 32078683
- [Background] Burgos AM, Saver JL. Evidence that Tenecteplase Is Noninferior to Alteplase for Acute Ischemic Stroke: Meta-Analysis of 5 Randomized Trials. Stroke. 2019 Aug;50(8):2156-2162. doi: 10.1161/STROKEAHA.119.025080. Epub 2019 Jul 18. PMID 31318627
- [Background] Hacke W, Kaste M, Bluhmki E, Brozman M, Davalos A, Guidetti D, Larrue V, Lees KR, Medeghri Z, Machnig T, Schneider D, von Kummer R, Wahlgren N, Toni D; ECASS Investigators. Thrombolysis with alteplase 3 to 4.5 hours after acute ischemic stroke. N Engl J Med. 2008 Sep 25;359(13):1317-29. doi: 10.1056/NEJMoa0804656. PMID 18815396
- [Background] Campbell BCV, Ma H, Ringleb PA, Parsons MW, Churilov L, Bendszus M, Levi CR, Hsu C, Kleinig TJ, Fatar M, Leys D, Molina C, Wijeratne T, Curtze S, Dewey HM, Barber PA, Butcher KS, De Silva DA, Bladin CF, Yassi N, Pfaff JAR, Sharma G, Bivard A, Desmond PM, Schwab S, Schellinger PD, Yan B, Mitchell PJ, Serena J, Toni D, Thijs V, Hacke W, Davis SM, Donnan GA; EXTEND, ECASS-4, and EPITHET Investigators. Extending thrombolysis to 4.5-9 h and wake-up stroke using perfusion imaging: a systematic review and meta-analysis of individual patient data. Lancet. 2019 Jul 13;394(10193):139-147. doi: 10.1016/S0140-6736(19)31053-0. Epub 2019 May 22. PMID 31128925
- [Background] Emberson J, Lees KR, Lyden P, Blackwell L, Albers G, Bluhmki E, Brott T, Cohen G, Davis S, Donnan G, Grotta J, Howard G, Kaste M, Koga M, von Kummer R, Lansberg M, Lindley RI, Murray G, Olivot JM, Parsons M, Tilley B, Toni D, Toyoda K, Wahlgren N, Wardlaw J, Whiteley W, del Zoppo GJ, Baigent C, Sandercock P, Hacke W; Stroke Thrombolysis Trialists' Collaborative Group. Effect of treatment delay, age, and stroke severity on the effects of intravenous thrombolysis with alteplase for acute ischaemic stroke: a meta-analysis of individual patient data from randomised trials. Lancet. 2014 Nov 29;384(9958):1929-35. doi: 10.1016/S0140-6736(14)60584-5. Epub 2014 Aug 5. PMID 25106063
- [Background] Kunz WG, Hunink MG, Almekhlafi MA, Menon BK, Saver JL, Dippel DWJ, Majoie CBLM, Jovin TG, Davalos A, Bracard S, Guillemin F, Campbell BCV, Mitchell PJ, White P, Muir KW, Brown S, Demchuk AM, Hill MD, Goyal M; HERMES Collaborators. Public health and cost consequences of time delays to thrombectomy for acute ischemic stroke. Neurology. 2020 Nov 3;95(18):e2465-e2475. doi: 10.1212/WNL.0000000000010867. Epub 2020 Sep 17. PMID 32943483
- [Background] Huang X, Cheripelli BK, Lloyd SM, Kalladka D, Moreton FC, Siddiqui A, Ford I, Muir KW. Alteplase versus tenecteplase for thrombolysis after ischaemic stroke (ATTEST): a phase 2, randomised, open-label, blinded endpoint study. Lancet Neurol. 2015 Apr;14(4):368-76. doi: 10.1016/S1474-4422(15)70017-7. Epub 2015 Feb 26. PMID 25726502
- [Background] Logallo N, Novotny V, Assmus J, Kvistad CE, Alteheld L, Ronning OM, Thommessen B, Amthor KF, Ihle-Hansen H, Kurz M, Tobro H, Kaur K, Stankiewicz M, Carlsson M, Morsund A, Idicula T, Aamodt AH, Lund C, Naess H, Waje-Andreassen U, Thomassen L. Tenecteplase versus alteplase for management of acute ischaemic stroke (NOR-TEST): a phase 3, randomised, open-label, blinded endpoint trial. Lancet Neurol. 2017 Oct;16(10):781-788. doi: 10.1016/S1474-4422(17)30253-3. Epub 2017 Aug 2. PMID 28780236
- [Background] Kheiri B, Osman M, Abdalla A, Haykal T, Ahmed S, Hassan M, Bachuwa G, Al Qasmi M, Bhatt DL. Tenecteplase versus alteplase for management of acute ischemic stroke: a pairwise and network meta-analysis of randomized clinical trials. J Thromb Thrombolysis. 2018 Nov;46(4):440-450. doi: 10.1007/s11239-018-1721-3. PMID 30117036
- [Result] Warner JJ, Harrington RA, Sacco RL, Elkind MSV. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke. Stroke. 2019 Dec;50(12):3331-3332. doi: 10.1161/STROKEAHA.119.027708. Epub 2019 Oct 30. No abstract available. PMID 31662117
- [Result] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Result] Liu L, Chen W, Zhou H, Duan W, Li S, Huo X, Xu W, Huang L, Zheng H, Liu J, Liu H, Wei Y, Xu J, Wang Y; Chinese Stroke Association Stroke Council Guideline Writing Committee. Chinese Stroke Association guidelines for clinical management of cerebrovascular disorders: executive summary and 2019 update of clinical management of ischaemic cerebrovascular diseases. Stroke Vasc Neurol. 2020 Jun;5(2):159-176. doi: 10.1136/svn-2020-000378. Epub 2020 Jun 18. PMID 32561535
- [Result] Ma H, Campbell BCV, Parsons MW, Churilov L, Levi CR, Hsu C, Kleinig TJ, Wijeratne T, Curtze S, Dewey HM, Miteff F, Tsai CH, Lee JT, Phan TG, Mahant N, Sun MC, Krause M, Sturm J, Grimley R, Chen CH, Hu CJ, Wong AA, Field D, Sun Y, Barber PA, Sabet A, Jannes J, Jeng JS, Clissold B, Markus R, Lin CH, Lien LM, Bladin CF, Christensen S, Yassi N, Sharma G, Bivard A, Desmond PM, Yan B, Mitchell PJ, Thijs V, Carey L, Meretoja A, Davis SM, Donnan GA; EXTEND Investigators. Thrombolysis Guided by Perfusion Imaging up to 9 Hours after Onset of Stroke. N Engl J Med. 2019 May 9;380(19):1795-1803. doi: 10.1056/NEJMoa1813046. PMID 31067369
- [Result] Thomalla G, Simonsen CZ, Boutitie F, Andersen G, Berthezene Y, Cheng B, Cheripelli B, Cho TH, Fazekas F, Fiehler J, Ford I, Galinovic I, Gellissen S, Golsari A, Gregori J, Gunther M, Guibernau J, Hausler KG, Hennerici M, Kemmling A, Marstrand J, Modrau B, Neeb L, Perez de la Ossa N, Puig J, Ringleb P, Roy P, Scheel E, Schonewille W, Serena J, Sunaert S, Villringer K, Wouters A, Thijs V, Ebinger M, Endres M, Fiebach JB, Lemmens R, Muir KW, Nighoghossian N, Pedraza S, Gerloff C; WAKE-UP Investigators. MRI-Guided Thrombolysis for Stroke with Unknown Time of Onset. N Engl J Med. 2018 Aug 16;379(7):611-622. doi: 10.1056/NEJMoa1804355. Epub 2018 May 16. PMID 29766770
- [Result] Seners P, Turc G, Maier B, Mas JL, Oppenheim C, Baron JC. Incidence and Predictors of Early Recanalization After Intravenous Thrombolysis: A Systematic Review and Meta-Analysis. Stroke. 2016 Sep;47(9):2409-12. doi: 10.1161/STROKEAHA.116.014181. Epub 2016 Jul 26. PMID 27462117
- [Result] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Result] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Result] Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GW, Cognard C, Cohen DJ, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Baxter BW, Devlin TG, Lopes DK, Reddy VK, du Mesnil de Rochemont R, Singer OC, Jahan R; SWIFT PRIME Investigators. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. N Engl J Med. 2015 Jun 11;372(24):2285-95. doi: 10.1056/NEJMoa1415061. Epub 2015 Apr 17. PMID 25882376
- [Result] Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama a Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 2015 Jan 1;372(1):11-20. doi: 10.1056/NEJMoa1411587. Epub 2014 Dec 17. PMID 25517348
- [Result] Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 2015 Mar 12;372(11):1009-18. doi: 10.1056/NEJMoa1414792. Epub 2015 Feb 11. PMID 25671797
- [Result] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Result] Fassbender K, Walter S, Grunwald IQ, Merzou F, Mathur S, Lesmeister M, Liu Y, Bertsch T, Grotta JC. Prehospital stroke management in the thrombectomy era. Lancet Neurol. 2020 Jul;19(7):601-610. doi: 10.1016/S1474-4422(20)30102-2. PMID 32562685
- [Result] Bivard A, Lin L, Parsonsb MW. Review of stroke thrombolytics. J Stroke. 2013 May;15(2):90-8. doi: 10.5853/jos.2013.15.2.90. Epub 2013 May 31. PMID 24324944
- [Result] Parsons M, Spratt N, Bivard A, Campbell B, Chung K, Miteff F, O'Brien B, Bladin C, McElduff P, Allen C, Bateman G, Donnan G, Davis S, Levi C. A randomized trial of tenecteplase versus alteplase for acute ischemic stroke. N Engl J Med. 2012 Mar 22;366(12):1099-107. doi: 10.1056/NEJMoa1109842. PMID 22435369
- [Result] Coutts SB, Dubuc V, Mandzia J, Kenney C, Demchuk AM, Smith EE, Subramaniam S, Goyal M, Patil S, Menon BK, Barber PA, Dowlatshahi D, Field T, Asdaghi N, Camden MC, Hill MD; TEMPO-1 Investigators. Tenecteplase-tissue-type plasminogen activator evaluation for minor ischemic stroke with proven occlusion. Stroke. 2015 Mar;46(3):769-74. doi: 10.1161/STROKEAHA.114.008504. Epub 2015 Feb 12. PMID 25677596
- [Result] Campbell BCV, Mitchell PJ, Churilov L, Yassi N, Kleinig TJ, Dowling RJ, Yan B, Bush SJ, Dewey HM, Thijs V, Scroop R, Simpson M, Brooks M, Asadi H, Wu TY, Shah DG, Wijeratne T, Ang T, Miteff F, Levi CR, Rodrigues E, Zhao H, Salvaris P, Garcia-Esperon C, Bailey P, Rice H, de Villiers L, Brown H, Redmond K, Leggett D, Fink JN, Collecutt W, Wong AA, Muller C, Coulthard A, Mitchell K, Clouston J, Mahady K, Field D, Ma H, Phan TG, Chong W, Chandra RV, Slater LA, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Bladin CF, Sharma G, Desmond PM, Parsons MW, Donnan GA, Davis SM; EXTEND-IA TNK Investigators. Tenecteplase versus Alteplase before Thrombectomy for Ischemic Stroke. N Engl J Med. 2018 Apr 26;378(17):1573-1582. doi: 10.1056/NEJMoa1716405. PMID 29694815
- [Derived] Liu H, Jin A, Pan Y, Meng X, Li H, Li Z, Wang Y, Li S. Efficacy and Safety of Intravenous Tenecteplase Versus Alteplase in Treating Acute Ischemic Stroke With Diabetes and Admission Hyperglycemia. J Am Heart Assoc. 2024 Oct 15;13(20):e036393. doi: 10.1161/JAHA.124.036393. Epub 2024 Oct 11. PMID 39392168
- [Derived] Wang Y, Li S, Pan Y, Li H, Parsons MW, Campbell BCV, Schwamm LH, Fisher M, Che F, Dai H, Li D, Li R, Wang J, Wang Y, Zhao X, Li Z, Zheng H, Xiong Y, Meng X; TRACE-2 Investigators. Tenecteplase versus alteplase in acute ischaemic cerebrovascular events (TRACE-2): a phase 3, multicentre, open-label, randomised controlled, non-inferiority trial. Lancet. 2023 Feb 25;401(10377):645-654. doi: 10.1016/S0140-6736(22)02600-9. Epub 2023 Feb 9. PMID 36774935
- [Derived] Li S, Campbell BCV, Schwamm LH, Fisher M, Parsons M, Li H, Pan Y, Wang Y; TRACE II investigators. Tenecteplase Reperfusion therapy in Acute ischaemic Cerebrovascular Events-II (TRACE II): rationale and design. Stroke Vasc Neurol. 2022 Feb;7(1):71-76. doi: 10.1136/svn-2021-001074. Epub 2021 Aug 26. PMID 34446531